CLINICAL TRIAL: NCT04163640
Title: Ovarian Rejuvenation Through Intra-ovarian Injection of Platelet Rich Plasma for Women With Premature Ovarian Insufficiency (POI) and Poor Ovarian Response (POR)
Brief Title: Ovarian Rejuvenation for Premature Ovarian Insufficiency and Poor Ovarian Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMA-2019-05
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Failure; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to this group will receive the intra-ovarian platelet rich plasma injection
  Interventions: Other: intra-ovarian platelet rich plasma injection
- Control Group (No Intervention): Patients randomized to this group will not receive the intra-ovarian platelet rich plasma injection

INTERVENTIONS:
Other: intra-ovarian platelet rich plasma injection — patients will undergo a transvaginal intra-ovarian platelet rich plasma injection
  Arms: Intervention Group

SUMMARY:
The objective of this study is to perform a prospective randomized controlled trial seeking to characterize the effects of intra-ovarian injection of platelet rich plasma (PRP) on biomarkers of ovarian reserve as well as IVF outcomes in women with primary ovarian insufficiency (POI) and poor ovarian response (POR) who decline the use of an egg donor to establish a pregnancy.

DETAILED DESCRIPTION:
Patients will be randomized to either receive the intra-ovarian PRP injection procedure or not. Regardless of randomization patients will be re-assessed at the same time points for ovarian reserve parameters. If antral follicles are detected at follow up, patients will undergo controlled ovarian hyperstimulation and a routine in vitro fertilization cycle as per protocol.

ELIGIBILITY:
Inclusion criteria

1. POI according to ESHRE criteria (patient must fit both criteria):

   1. presence of menstrual disturbance defined as oligo/amenorrhea for at least 4 months
   2. biochemical confirmation as evidenced by an elevated FSH level >25 IU/L on two occasions > 4 weeks apart
2. POR defined by at least two prior cycles with POR (≤3 oocytes retrieved with a conventional stimulation protocol, or a cancelled cycle due to poor response)
3. Patients declining ovum donation treatment

Exclusion criteria

1. Age <18yo or >38yrs
2. Autoimmune or sex chromosome etiology of POI
3. Ongoing malignancy
4. Previous ovarian surgery
5. Previous gonadotoxic treatment
6. Anticoagulant use for which plasma infusion is contraindicated
7. FMR1 mutations
8. If the duration of the amenorrhea is more than 2 years, patients are discouraged to participate, although it is not an exclusion criterion.
9. Patients with only 1 ovary
10. BMI > 35
11. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
12. Surgically obtained sperm
13. Presence of hydrosalpinges that communicate with endometrial cavity
14. Single gene disorder or chromosomal rearrangement requiring a more detailed embryonic genetic analysis
15. Diagnosis of endometrial insufficiency: prior cycle with maximal endometrial thickness ≤ 6mm, abnormal endometrial pattern (failure to attain a trilaminar appearance), persistent endometrial fluid
16. Use of a gestational carrier
17. Any contraindications to undergoing in vitro fertilization or gonadotropin stimulation
18. Known ovaries that are not accessible transvaginally.
19. Ovarian endometrioma(s) or dermoid cyst(s) identified via transvaginal ultrasound
20. FSH > 40iu/l

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
number of participants with a mature oocyte retrieved- POI group | 24 hours post egg retrieval procedure
  success or failure is determined by the retrieval of at least one mature oocyte
number of mature oocytes retrieved- POR group | 24 hours post egg retrieval procedure
  the total number of mature oocytes retrieved

CONTACTS AND LOCATIONS:
Overall Officials: Emre U Seli, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (2):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herlihy NS, Cakiroglu Y, Whitehead C, Reig A, Tiras B, Scott RT Jr, Seli E. Effect of intraovarian platelet-rich plasma injection on IVF outcomes in women with poor ovarian response: the PROVA randomized controlled trial. Hum Reprod. 2024 May 9:deae093. doi: 10.1093/humrep/deae093. Online ahead of print. PMID 38725194